CLINICAL TRIAL: NCT01762631
Title: Baby Bottle: Remote Food Photography Method in Infants
Brief Title: Remote Food Photography Method in Infants
Acronym: BabyBottle
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 12035
Record Dates: First submitted 2012-12-17; First posted 2013-01-08 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Estimating Infant Food Intake

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: All participants enrolled between November 2012 and March 2013 under the original protocol.
- Cohort 2: After Cohort 1 was completed, the study investigators changed the protocol to eliminate the photograph/weight of the powdered formula alone in each bottle to reduce burden. All other protocol procedures remained the same. Cohort 2 participants enrolled between April 2013 and May 2014.

SUMMARY:
The purpose of this study is to determine if digital photography on a Smartphone and the Remote Food Photography Method (RFPM) can estimate infant formula intake. This is a validation study; there is no hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Willing to complete 2 study visits at Pennington Biomedical (PBRC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 75 men and women will be recruited to participate in a 2-week pilot study involving infant formula preparation. Participation is open to all adult individuals.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center; Corby Martin, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- See also: PBRC Website description and webscreening link — http://www.pbrc.edu/clinical-trials/?studyid=151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited through advertisements and targeted emails directed to residents of the Greater Baton Rouge area.
Groups:
- Study Participants in Cohort 1; Study Participants in Cohort 2: No intervention, time frame of visit determined Cohort 1 vs Cohort 2
Period: Overall Study
Arm/Group | Study Participants in Cohort 1 | Study Participants in Cohort 2
Started | 53 | 22
Completed | 53 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adults who were caregivers or non-caregivers of infants
Groups:
- Study Participants In Cohort 1; Study Participants in Cohort 2: No intervention- time frame of visits determined Cohort 1 vs Cohort 2
- Total: Total of all reporting groups
Arm/Group | Study Participants In Cohort 1 | Study Participants in Cohort 2 | Total
Number analyzed (Participants) | 53 | 22 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (13.8) | 33.1 (11.9) | 32.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 20 | 67
  Male | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 53 | 22 | 75
Caregiver Status [Count of Participants; unit: Participants]
  Caregiver of Infant | 28 | 14 | 42
  Non-caregiver of Infant | 25 | 8 | 33

OUTCOME MEASURES:

1. Primary Outcome: Kilocalorie (Kcal) Difference Between Methods for All Prepared Bottles
Description: Kilocalorie (Kcal) Difference in prepared infant formula intake detected in a bottle between the Remote Food Photography Method (RFPM) and direct weighing
  Kilocalorie difference between the Remote Food Photography Method and direct weighing with all bottles that were prepared included
  Kilocalorie difference is Remote Food Photography Method - Direct Weighing
Time Frame: Measures will be performed twice about 5-10 days apart
Population: Since Cohort 2 had a modified protocol where the step involving photographs and direct weights of bottles with powdered formula only was not completed, the kilocalories for all participants in Cohort 2 cannot be determined. Powder not water is the source of kilocalories in formula; we could not accurately determine kilocalories without this step.
Measure: Mean (Standard Deviation); unit: kilocalories
Arm/Group | Study Participants in Cohort 1 | Study Participants in Cohort 2
Number analyzed (Participants) | 53 | 0
kilocalories
  Remote Food Photography Method | 82.1 (42.3) |
  Direct Weighing | 85.3 (43.2) |

2. Secondary Outcome: Kilocalorie (Kcal) Difference Between Different Bottle Sizes
Description: Kilocalorie difference between the Remote Food Photography Method and direct weighing separately analyzed by the four different bottle sizes that were prepared (2 oz bottles only, 4 oz bottles only, 6 oz bottles only, and 8 oz bottles only). Each participant prepared 3 sets of 2 oz bottles, 3 sets of 4 oz bottles, 3 sets of 6 oz bottles, and 3 sets of 8 oz bottles and all bottles of the specified size were included in the analysis.
  Kilocalorie difference is Remote Food Photography Method - Direct Weighing
Time Frame: Measures will be performed twice about 5-10 days apart
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilocalories
Arm/Group | Study Participants in Cohort 1 | Study Participants in Cohort 2
Number analyzed (Participants) | 53 | 0
kilocalories
  Remote Food Photography-2 oz prepared bottles | 34.2 (7.8) |
  Direct Weighing- 2 oz prepared bottles | 35.8 (7.6) |
  Remote Food Photography-4 oz prepared bottles | 64.5 (13.8) |
  Direct Weighing- 4 oz prepared bottles | 69.3 (16.8) |
  Remote Food Photography-6 oz prepared bottles | 94.9 (22.4) |
  Direct Weighing- 6 oz prepared bottles | 101.1 (25.3) |
  Remote Food Photography-8 oz prepared bottles | 135.0 (28.6) |
  Direct Weighing- 8 oz prepared bottles | 134.9 (32.8) |

3. Other Pre Specified Outcome: Gram Weight of Infant Formula Provision Between Participants Who Identified as Infant Caregivers and Infant Non-caregivers for 2 oz Prepared Bottles Only
Description: A caregiver will be defined as an individual who is a parent, grandparent, sibling, aunt or uncle, or nanny or babysitter who has provided care to an infant within the last 12 months.
  Gram weight by direct weighing comparing the caregivers and non-caregivers in infant formula provision (not simulated intake) in 2 oz prepared bottles only. Each participant prepared 3 sets of 2 oz bottles, and all bottles of the specified size were included in the analysis.
Time Frame: Measures will be performed twice about 5-10 days apart
Population: Number of participants' data analyzed is broken down between those who identified as infant caregivers and those who identified as infant non-caregivers.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Study Participants in Cohort 1 | Study Participants in Cohort 2
Number analyzed (Participants) | 53 | 22
grams
  Infant Caregivers: number analyzed (Participants) | 28 | 14
  Infant Caregivers | 57.5 (8.0) | 64.2 (6.7)
  Infant Non-caregivers: number analyzed (Participants) | 25 | 8
  Infant Non-caregivers | 57.8 (7.6) | 58.9 (11.5)

4. Other Pre Specified Outcome: Gram Weight of Infant Formula Provision Between Participants Who Identified as Infant Caregivers and Infant Non-caregivers for 4 oz Prepared Bottles Only
Description: A caregiver will be defined as an individual who is a parent, grandparent, sibling, aunt or uncle, or nanny or babysitter who has provided care to an infant within the last 12 months.
  Gram weight by direct weighing comparing the caregivers and non-caregivers in infant formula provision (not simulated intake) in 4 oz prepared bottles only. Each participant prepared 3 sets of 4 oz bottles, and all bottles of the specified size were included in the analysis.
Time Frame: Measures will be performed twice about 5-10 days apart
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Study Participants in Cohort 1 | Study Participants in Cohort 2
Number analyzed (Participants) | 53 | 22
grams
  Infant Caregivers: number analyzed (Participants) | 28 | 14
  Infant Caregivers | 115.0 (16.2) | 128.6 (13.7)
  Infant Non-caregivers: number analyzed (Participants) | 25 | 8
  Infant Non-caregivers | 115.4 (16.7) | 111.7 (16.6)

5. Other Pre Specified Outcome: Gram Weight of Infant Formula Provision Between Participants Who Identified as Infant Caregivers and Infant Non-caregivers for 6 oz Prepared Bottles Only
Description: A caregiver will be defined as an individual who is a parent, grandparent, sibling, aunt or uncle, or nanny or babysitter who has provided care to an infant within the last 12 months.
  Gram weight by direct weighing comparing the caregivers and non-caregivers in infant formula provision (not simulated intake) in 6 oz prepared bottles only. Each participant prepared 3 sets of 6 oz bottles, and all bottles of the specified size were included in the analysis.
Time Frame: Measures will be performed twice about 5-10 days apart
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Study Participants in Cohort 1 | Study Participants in Cohort 2
Number analyzed (Participants) | 53 | 22
grams
  Infant Caregivers: number analyzed (Participants) | 28 | 14
  Infant Caregivers | 176.6 (34.8) | 195.0 (19.5)
  Infant Non-caregivers: number analyzed (Participants) | 25 | 8
  Infant Non-caregivers | 180.7 (36.1) | 166.9 (25.9)

6. Other Pre Specified Outcome: Gram Weight of Infant Formula Provision Between Participants Who Identified as Infant Caregivers and Infant Non-caregivers for 8 oz Prepared Bottles Only
Description: A caregiver will be defined as an individual who is a parent, grandparent, sibling, aunt or uncle, or nanny or babysitter who has provided care to an infant within the last 12 months.
  Gram weight by direct weighing comparing the caregivers and non-caregivers in infant formula provision (not simulated intake) in 8 oz prepared bottles only. Each participant prepared 3 sets of 8 oz bottles, and all bottles of the specified size were included in the analysis.
Time Frame: Measures will be performed twice about 5-10 days apart
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Study Participants in Cohort 1 | Study Participants in Cohort 2
Number analyzed (Participants) | 53 | 22
grams
  Infant Caregivers: number analyzed (Participants) | 28 | 14
  Infant Caregivers | 244.3 (46.3) | 249.3 (24.1)
  Infant Non-caregivers: number analyzed (Participants) | 25 | 8
  Infant Non-caregivers | 243.8 (37.9) | 222.8 (27.9)

ADVERSE EVENTS:
Time Frame: The study time period was 5-10 days.
Description: In this study, an adverse event or experience is defined as any health-related unfavorable or unintended medical occurrence that happens after screening. We anticipate most adverse events will be mild and the participant will be able to resume activities within a day or two of reporting the event. Adverse Event reporting will follow the requirements of the Pennington Biomedical Research Center Institutional Review Board.
Arm/Group | Study Participants in Cohort 1 | Study Participants in Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/22
Other Adverse Events (participants affected / at risk) | 0/53 | 0/22

LIMITATIONS AND CAVEATS:
Without powder alone, kilocalories for all participants in Cohort 2 cannot be determined due to the protocol modification completed prior to Cohort 2. Therefore, primary and secondary outcome results cannot be determined for Cohort 2 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes